CLINICAL TRIAL: NCT05945784
Title: Exploring Accessible Beauty: A Study on Enhancing Beauty Product Accessibility for Individuals With Upper Extremity Deficits
Brief Title: Exploring Accessible Beauty for Individuals With Upper Extremity Deficits
Status: Completed | Type: Observational
Sponsor: Casa Colina Hospital and Centers for Healthcare (Other)
Responsible Party: Principal Investigator, Emily Rosario, Executive Director, Casa Colina Hospital and Centers for Healthcare
Other Study IDs: IRB: 000000001
Record Dates: First submitted 2023-06-27; First posted 2023-07-14 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic; Stroke (CVA) or TIA; Stroke, Acute; Traumatic Brain Injury; SCI - Spinal Cord Injury; Ehlers-Danlos Syndromes (EDS); Lupus Erythematosus; Guillain-Barre Syndrome; Multiple Sclerosis; Myasthenia Gravis; Amyotrophic Lateral Sclerosis; Graves Disease; Muscular Dystrophies
Keywords: upper extremity disabilities; limited mobility; dexterity impairments; muscle weakness
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Stroke; Brain Injuries, Traumatic; Spinal Cord Injuries; Ehlers-Danlos Syndrome; Guillain-Barre Syndrome; Multiple Sclerosis; Myasthenia Gravis; Amyotrophic Lateral Sclerosis; Graves Disease; Muscular Dystrophies; Muscle Weakness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Minimal to moderate upper extremity deficits: * Individuals aged 18 years to 55 years.
  * Minimal to moderate upper extremity deficits, including but not limited to limited mobility or dexterity impairments.
  * Regular users of beauty products.
  * Able to understand and communicate in the language of the study.
  Interventions: Other: Use of Rare Beauty makeup products

INTERVENTIONS:
Other: Use of Rare Beauty makeup products — Participants will be provided with a selection of beauty products items including foundation, concealer, blush, highlighter, and lipstick, specifically chosen for their potential accessibility features. They will have a specified trial period during which they can use the products as part of their regular beauty routines.

SUMMARY:
The purpose of this study is to investigate the accessibility of beauty products for individuals with upper extremity disabilities. By examining various factors such as packaging design, product applicators, and ease of use, this research aims to identify barriers faced by individuals with upper extremity disabilities or visual deficits when using beauty products. The study seeks to provide insights and recommendations for improving the accessibility of beauty products, ultimately promoting inclusivity and enhancing the overall beauty experience for individuals with disabilities.

DETAILED DESCRIPTION:
Individuals with upper extremity disabilities face unique challenges when it comes to using beauty products. These disabilities can include conditions such as limb loss, limited mobility, or dexterity impairments, which can significantly impact their ability to engage in self-care and beauty routines. The accessibility of beauty products is crucial to ensure that individuals with upper extremity disabilities have equal opportunities to participate in activities that promote self-expression and confidence.

Research in the field of accessible design has highlighted the importance of inclusive product development across various industries, including cosmetics and personal care. However, limited attention has been given specifically to beauty products and their usability for individuals with upper extremity disabilities.

To address this gap, studies are being conducted to assess the accessibility of beauty products and identify potential barriers and solutions. These studies typically examine factors such as packaging design, ergonomics of product applicators, ease of grip, and maneuverability. By understanding the specific challenges faced by individuals with upper extremity disabilities, researchers can propose modifications and design considerations that enhance accessibility.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged 18 years to 55 years.

* Minimal to moderate upper extremity deficits, including but not limited to limited mobility or dexterity impairments.
* Regular users beauty products.
* Able to understand and communicate in the language of the study.

Exclusion Criteria:

* Individuals below 18 years of age or over the age of 55.
* Individuals without upper extremity deficits or with severe upper extremity deficits that may affect the participant's ability to engage in study activities.
* Participants who are not regular users of beauty products.
* Inability to understand and communicate in the language of the study.
* Any medical or psychological condition that may affect the participant's ability to provide informed consent or engage in the study activities safely.
* Individuals who experience facial skin or eye irritation reported by subject or observed by evaluator at baseline visit
* History of allergic reactions, and/or known allergies to cosmetic ingredients, toiletries, sunscreens, etc.
* Immunocompromised subjects
* Individuals who may experience changes in hormones, such as just those using oral contraception for less than three months before the screening visit or who have changed hormonal contraceptive methods within the three months before the Baseline visit or planning to modify hormonal contraception treatment within the duration of the study.
* Known to be pregnant, lactating or planning to become pregnant within six months. Subjects who become pregnant during the study must inform the Principal Investigator immediately.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A convenience sample of individuals aged 18 and above, with upper extremity deficits, will be recruited for this study. Efforts will be made to include participants with a range of upper extremity deficits and experiences with beauty products.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Likert Scale | Complete on Day 7
  It is a validated self-reported instrument to assess packaging of the makeup. A few questions will focus on shape of the cap, length of the wand, shape of the doe foot, finish of the components, how it affects grip, and weight of the component/applicator. Possible scores range from 1 (strongly disagree) to 5 (strongly agree).
Likert Scale | Complete on Day 14
  It is a validated self-reported instrument to assess packaging of the makeup. A few questions will focus on shape of the cap, length of the wand, shape of the doe foot, finish of the components, how it affects grip, and weight of the component/applicator. Possible scores range from 1 (strongly disagree) to 5 (strongly agree).
Pre-test Questionnaire | At baseline
  Participants will complete questionnaires that assess their demographics, disability characteristics, and previous experiences with beauty products.
Accessibility Evaluation | Day 7, after use of beauty products
  Participants will evaluate the beauty products based on predefined criteria, including ease of grip, maneuverability, packaging design, and product applicators. They will document their experiences, challenges faced, and any suggestions for improvements. Possible scores range from 1 (strongly disagree) to 5 (strongly agree).
Accessibility Evaluation | Day 14, after use of beauty products at end of study
  Participants will evaluate the beauty products based on predefined criteria, including ease of grip, maneuverability, packaging design, and product applicators. They will document their experiences, challenges faced, and any suggestions for improvements. Possible scores range from 1 (strongly disagree) to 5 (strongly agree).
Post-test Questionnaire | Day 14, after use of beauty products at end of study
  Participants will assess changes in their perceptions and experiences with the beauty products. This will include questions about satisfaction, usability, and any perceived improvements in accessibility. Possible scores range from 1 (strongly disagree) to 5 (strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Emily Rosario, PhD, Principal Investigator — Casa Colina Hospital and Centers for Healthcare
Locations (1):
- Casa Colina Hospital and Centers for Healthcare, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skelton H, Gill S, Al Zidjaly N, et al. Exploring the Accessibility of Beauty Products for Individuals with Mobility Disabilities. J Appl Cosmetol. 2020;38(3):65-72.
- [Background] Smith A, Johnson R, Thompson A, et al. Enhancing Accessibility: Designing Inclusive Beauty Products for All Abilities. J Inclusive Design. 2021;1(2):89-102
- [Background] Chen L, Kim D, Park J, et al. A Review on Product Accessibility Evaluation Methods for People with Disabilities. Int J Ind Ergon. 2019;71:103-117. doi:10.1016/j.ergon.2018.11.007